CLINICAL TRIAL: NCT06576453
Title: Mixed-method Evaluation of a Parental Psychoeducation Programme in a Suicide Risk Prevention Group
Acronym: Pepps_Mix
Status: Recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP231318
Record Dates: First submitted 2024-07-04; First posted 2024-08-28 (Actual); Last update posted 2024-08-28 (Actual); Status verified 2024-08

CONDITIONS: Suicide Prevention
MeSH Terms: conditions — Suicide Prevention

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- All of the participants: Parents participate in the PEPPS program (Parental psychoeducation program for suicide risk prevention) This is a group family psychoeducation program for parents child under 15 years 6 months having been urgently assessed at Robert University Hospital discharged for suicidal ideation or attempted suicide.
  This program is built according to a global model based on:
  * A support program for parents of Resourceful adolescents: parent of adolescents support program not specific to the theme of suicidal risk taking place in 3 to 4 sessions of 2 hours.
  * The global program of the Suicide Prevention Intervention Center at the Children Hospital of Philadelphia which offers a multi-family group intervention (parents and children).
  * The recommendations of the High Authority of Health which recommend an intervention psychoeducation type.
  Interventions: Behavioral: Self-questionnaire WHOQOL-bref; Behavioral: Self-questionnaire Evaluation Inventory - Parent; Behavioral: quiz of knowledge
- Participants - qualitative interview: Semi-structured interviews (qualitative) will be carried out with parents who have followed either all or part of the sessions of the band. The parents interviewed will be chosen based on the wealth of information they will be likely to contribute to the study.The sampling method will follow the "snowball" model, described by Kathy Charmaz. According to this, the characteristics of new participants will be determined according to the results of the analysis of the first interviews until data saturation. We will conclude with the latter when no new information emerges from the data collection.
  Interventions: Behavioral: Self-questionnaire WHOQOL-bref; Behavioral: Self-questionnaire Evaluation Inventory - Parent; Behavioral: quiz of knowledge; Behavioral: semi-structured interviews (qualitative)

INTERVENTIONS:
Behavioral: Self-questionnaire WHOQOL-bref — Parents must complete the self-questionnaire WHOQOL-bref after the first and the last session of the Pepps program.
Behavioral: Self-questionnaire Evaluation Inventory - Parent — Parents must complete the self-questionnaire Evaluation Inventory - Parent after the last session of the Pepps program.
Behavioral: quiz of knowledge — Parents must complete the quiz of knowledge after the first and the last session of the Pepps program.
Behavioral: semi-structured interviews (qualitative) — In the month following the last session of the program, the semi-structured interviews (qualitative) will be carried out with parents who have followed either all or part of the sessions of the band.
  Groups: Participants - qualitative interview

SUMMARY:
The number of emergency consultations for children and adolescents for suicidal ideation and suicide attempts has been rising steadily since 2010, and even more so since 2020. In addition, 30% of children and adolescents who have committed a suicidal act reoffend within the year.

Psycho-education programmes for patients have been shown to be effective in a large number of psychiatric pathologies. The programs of psychoeducation for the caregivers of these patients have them also shown their effectiveness, however to date there is no parental psychoeducation program group, for the prevention of the suicidal risk of children and adolescents, which is validated. The service of child psychiatry at the Robert Debré hospital built a program for this purpose, according to current data from the science and has been offering it for 6 months to parents of patients who consulted for suicidal ideation. Rate this program through the description of its implementation would allow it to be validated, this in a dissemination objective. This validation through a mixed method would also allow us to describe the experience participants in this program and to understand improvements Track.

DETAILED DESCRIPTION:
Implementation study: non-randomized, single-center, quasi-experimental study before - after for the evaluation criteria of intermediate effectiveness (effectiveness). Study mixed qualitative-quantitative method for the evaluation of several judgment criteria.

The main objectives is to Evaluate the implementation of a parental psychoeducation program in a group of suicide prevention through parental support for the entire program.

The secondary objectives are to evaluate:

* reaching the target population (Reach)
* the intermediate effectiveness of the program
* the adoption of the program by health professionals
* the implementation on other dimensions
* the sustainability of the program

ELIGIBILITY:
Inclusion Criteria:

* Parent committing to participate in the 4 sessions of the parental psychoeducation prevention program suicide risk (PEPPS program)
* Parents of children under 15 years and 6 months
* Parents fluent in French

Exclusion Criteria:

* Lack of affiliation with a social security scheme or CMU (universal health coverage)
* Parents under guardianship or curatorship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Parents of a child under 15 years 6 months old urgently consulted at the Robert Debré hospital for ideas suicidal or attempted suicide
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2024-05-23 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
implementation of a program parental psychoeducation in prevention groups suicide (program PEPPS). | Week 5
  program membership = Number of parents who have been present at the 4 sessions / Number of parents included (having agreed to participate in the program)

SECONDARY OUTCOMES:
reaching the target population | Week 5
  number of parents to whom the program has been proposed / number of parents having had a child having consulted for suicidal ideation
Intermediate program effectiveness by comparison of levels of parents' responses between the start of program and the end of the last session of the program | Week 5
  level of knowledge about suicidal behavior: degree of certainty a knowledge quiz built for the program
Intermediate program effectiveness by comparison of levels of parents' responses between the start of program and the end of the last session of the program | Week 5
  parents' quality of life: score WHOQOL-BREF scale
adoption of the program by health professionals | Week 5
  number of emergency professionals offering program for parents / number of emergency professionals treating children having consulted for suicidal ideation
Implementation on other dimensions | Week 5
  Number of parents participating in at least a session
Implementation on other dimensions | Week 5
  Satisfaction of participating parents: Parent Evaluation self-questionnaire Inventory-Parent Treatment
Implementation on other dimensions | Week 5
  Describe the parents' experience participant in the PEPPS program: analysis qualitative (interview)
sustainability of the program (Maintenance): Interview | Week 9
  Identify the brakes and levers implementation of the program, in order to identify avenues for improvement and dissemination of psychoeducation program: analysis qualitative

CONTACTS AND LOCATIONS:
Locations (1):
- Robert Debré Hospital, Child and adolescent psychiatry department, Paris, Île-de-France Region, France